CLINICAL TRIAL: NCT01619306
Title: Knowledge and Attitudes of Patients and Healthcare Professionals on a Spectrum of Genetic Tests Relevant to Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/00752
Record Dates: First submitted 2012-04-02; First posted 2012-06-14 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objectives:

Primary objectives:

• The investigators aim to conduct a questionnaire survey in a South-East Asian tertiary institution, to assess whether breast cancer patients and their physicians would consider the use of three different kinds of genetic tests currently available to breast cancer patients:

* BRCA1/2 germline testing,
* CYP2D6 genotyping and
* Oncotype DX® testing.

Secondary objectives:

To explore factors which might influence their decisions on genetic testing, including:

1. Acceptability of the tests and anti-cancer management based on the test results
2. Reliability and affordability of the test
3. Ability of the test to influence treatment decisions
4. Broader implications of the test, e.g., psychosocial, financial impact Study design: Cross-sectional study, Survey Questionnaires were developed for 3 categories of individuals:

   * Patients with early stage breast cancer
   * Healthcare professionals caring for breast cancer patients
   * Medical students /cancer researchers The questionnaires for patients and medical students/cancer researchers are similar. The questionnaires contain a brief section on demographic information, interest in and past experience with genetic testing. Three hypothetical situations are described to determine if participants will agree to BRCA1/2 testing, CYP2D6 genotyping and Oncotype DX® testing, respectively. 18 categorical 'yes'/ 'no' questions explore reasons for their decisions. Each scenario requires a short, hand-written response.

The questionnaire for healthcare professionals contains a brief section on demographics and past experience with genetic testing. Three hypothetical situations are described to determine if healthcare professionals will recommend their patients for BRCA1/2 testing, CYP2D6 genotyping and Oncotype DX® testing, respectively. 12 categorical questions explore the reasons for their decision, and physicians are required to rank these in order of importance.

Distribution of questionnaires:

Questionnaires will be handed out to agreeable participants on the following occasions:

1. Patients- National University Health System Cancer Centre Level 3 amp; 4 waiting areas
2. Medical students - before or after lectures, or at personal contact
3. Cancer researchers - before or after lectures, or at personal contact
4. Healthcare professionals - before or after NUHS breast tumour board, or at personal contact Due caution will be exercised to ensure that the questionnaire is only handed out to subjects who are aged 21 years and above.

No subject identity will be collected for these questionnaires.

Rationale and Hypothesis:

BRCA1/2 germline testing, CYP2D6 genotyping and Oncotype DX® testing have all been approved for use in clinical practice, but controversy still exists surrounding their utility, and apart from BRCA1/2 mutation testing in high-risk individuals, genetic tests are not routinely performed in Singapore. BRCA1/2 germline mutation testing is performed in individuals at high risk for hereditary cancer. CYP2D6 genotype testing predicts the benefit of adjuvant tamoxifen therapy; poor and intermediate metabolisers of tamoxifen may have a higher risk of breast cancer recurrence due to lower efficacy of tamoxifen because of less efficient conversion of tamoxifen to endoxifen, the active metabolite of tamoxifen. Oncotype DX® testing is a gene-expression profiling test performed on a formalin-fixed paraffin embedded tumour specimen, to predict the risk of breast cancer recurrence and guide decisions on adjuvant chemotherapy. Understanding the attitudes of patients and medical professionals toward these genetic tests may help to guide medical oncologists in their clinical recommendations and utilization of these tests in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early stage breast cancer
* Healthcare professionals caring for breast cancer patients
* Medical students /cancer researchers

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Questionnaires will be handed out to agreeable participants on the following occasions. 1. Patients- National University Health System Cancer Centre Level 3 amp; 4 waiting areas 2. Medical students - before or after lectures, or at personal contact 3. Cancer researchers - before or after lectures, or at personal contact 4. Healthcare professionals - before or after NUHS breast tumour board, or at personal contact Due caution will be exercised to ensure that the questionnaire is only handed out to subjects who are aged 21 years and above.
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Conduct a questionnaire survey in a South-East Asian tertiary institution
  The investigators aim to conduct a questionnaire survey in a South-East Asian tertiary institution, to assess whether breast cancer patients and their physicians would consider the use of three different kinds of genetic tests currently available to breast cancer patients: BRCA1/2 germline testing, CYP2D6 genotyping and Oncotype DX® testing.

SECONDARY OUTCOMES:
To explore factors which might influence their decisions on genetic testing
  To explore factors which might influence their decisions on genetic testing, including:
  1. Acceptability of the tests and anti-cancer management based on the test results
  2. Reliability and affordability of the test
  3. Ability of the test to influence treatment decisions
  4. Broader implications of the test, e.g., psychosocial, financial impact

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore